CLINICAL TRIAL: NCT04463160
Title: Study of the Factors Favoring the Transition From Prediabetes to Diabetes on Reunion Island. Impact of the "Say No to Diabetes" Intervention.
Brief Title: Study of the Factors Favoring the Transition From Prediabetes to Diabetes on Reunion Island.
Acronym: PREDIABRUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2018/CHU/06; 2018-A03106-49 (Other: ID-RCB)
Record Dates: First submitted 2020-06-30; First posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prevention program for prediabetes "Say No to Diabetes" (Experimental)
  Interventions: Other: prevention program for prediabetes "Say No to Diabetes"
- No prevention program (No Intervention)

INTERVENTIONS:
Other: prevention program for prediabetes "Say No to Diabetes" — 10 therapeutic education sessions
  Arms: prevention program for prediabetes "Say No to Diabetes"

SUMMARY:
The management of diabetes and its complications in Reunion island is one of the priority areas of health. Indeed, the impact of diabetes on the health of the Reunion island population is major: the prevalence of diabetes treated in Reunion island is the highest in France (10% of the population), and gestational diabetes is found in 10% of pregnancies. Reunionese diabetics develop severe complications, in particular cardiovascular (strokes, myocardial infarction).

This results in 3 times higher mortality linked to diabetes on Reunion Island, in particular among those under 65 years of age. Despite all the screening and prevention programs put in place, the weight of diabetic disease continues to increase in our island, and this is more accelerated than in the other French departments with 4,300 new cases of diabetes / year, 95% of which type 2 diabetics (T2D). The presentation of type 2 diabetic patients in Reunion island also differs from the Metropolis with subjects more often female (56%), thinner and younger at the discovery of diabetes. These data highlight the need to better understand the factors underlying the diabetes "epidemic" in Reunion island.

The rise in blood sugar until the onset of diabetes is a continuous phenomenon reflecting the progressive suffering of the organs used to maintain carbohydrate homeostasis. Thus, we talk about fasting hyperglycemia when the fasting blood sugar is between 1.10 and 1.25 g / L (6.1-6.9 mmol / l) and glucose intolerance when the blood sugar 2 hours after taking 75 g of glucose is between 1.40 and 1.99 g / L (7.8-11.0 mmol / l). Subjects with fasting hyperglycemia or glucose intolerance constitute the target population at very high risk of developing diabetes (up to 70% of these subjects). They have an increased risk of developing diabetes at 1 year multiplied by 5 to 10 compared to normoglycemic subjects, hence the name "prediabetic subjects". This great variability in the risk of developing diabetes highlights the presence of associated risk / protective factors which it is important to find in order to adapt the monitoring and management. It is important in Reunion island, in view of the specificities presented by our population, to understand the pre-diabetes / diabetes transition and the risk and protective factors.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 25 to 70 with pre-diabetes defined by fasting blood sugar between 1.10 and 1.25 g / l (6.1 and 6.9 mmol / l) or blood sugar between 1.40 and 1.99 g / l (7.8 and 11.0 mmol / l) 2 hours after taking 75g of glucose (HGPO test), dating from less than 3 months.
* Consulting one of the general practitioners involved in the study, whatever the initial reason for the consultation
* able to answer a telephone survey questionnaire
* who have never been diagnosed or treated for diabetes with the exception of gestational diabetes
* Person affiliated or beneficiary of a social security scheme.
* Free, informed and written consent signed

Exclusion Criteria:

* People likely to leave Reunion within 2 years
* Persons placed under guardianship, curators, safeguard of justice, person participating in another research including an exclusion period still in progress.
* Person with severely impaired physical and / or psychological health, who, according to the investigator, may affect the compliance of the study participant.
* Pregnancy in progress

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-18 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The impact of the "Say No to Diabetes" intervention on the incidence of type 2 diabetes | 2 years
  Diabetes : fasting blood glucose ≥ 1.26 g / l (7 mmol / l), or blood sugar 2 hours after taking 75 g of glucose during HGPO ≥2 g / l (11.1 mmol / l)

SECONDARY OUTCOMES:
Numer of patients with diagnosic of type 2 diabetes in subjects identified as pre-diabetic | 2 years
  Prediabetes : fasting blood sugar is between 1.10 and 1.25 g / l (6.1 and 6.9 mmol / l) or a blood sugar level is between 1.40 and 1.99 g / l (7.8 and 11 0.0 mmol / l) 2 hours after taking 75g of glucose (HGPO test) Diabetes : fasting blood glucose ≥ 1.26 g / l (7 mmol / l), or blood sugar 2 hours after taking 75 g of glucose during HGPO ≥2 g / l (11.1 mmol / l)
Number of patients return to normal blood sugar | 2 years
  Normal blood sugar : fasting blood glucose <1.10 g / l (6.1mmol / l), or blood sugar 2 hours after taking 75 g of glucose during HGPO <1.40g / l (7.8 mmol / l).
HbA1c assay for the diagnosis of glucose intolerance and prediabetes compared to HGPO | 2 years
  HbA1c assay

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de la Réunion, Saint-Pierre, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anthony N, Bruneau L, Leruste S, Franco JM, Domercq A, Kowalczyk C, Nobecourt E, Marimoutou C. Diabetes incidence in subjects with PREDIABetes from ReUNion Island: the PREDIABRUN observational cohort study protocol. BMJ Open. 2022 Nov 21;12(11):e062520. doi: 10.1136/bmjopen-2022-062520. PMID 36410808